CLINICAL TRIAL: NCT04279145
Title: Evaluation of Echocardiographic Indices and Blood Biomarkers in Group 1 Pulmonary Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Moustafa Hosny Abdelmegeed Aly, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: group 1 PH
Record Dates: First submitted 2020-02-09; First posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Echocardiography

STUDY DESIGN:
Intervention Model Description: patients with primary pulmonary hypertension will submitted to : swanganz cath. detailed echocadiography blood samples for bio markers
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pulmonary hypertension group 1 (Experimental): each patient will be submitted to : swan-ganze catheterization detailed echocardiography blood sample for biomarkers (troponin, uric acid and micro RNA)
  Interventions: Device: swan ganze catheter /echocardiography

INTERVENTIONS:
Device: swan ganze catheter /echocardiography — Right heart catheterization and mixed venous blood samples will be obtained for ABG, biomarkers (troponin , uric acid and micro RNA).
  Each subject will have echocardiography, 6 MWD, clinical functional class and blood sample at the day of right heart catheterization or at least less than week of right heart catheterization

SUMMARY:
* To evaluate different echocardiographic indices in diagnosis and follow up of group 1 pulmonary hypertension.
* To evaluate blood biomarkers (troponin, uric acid and micro RNA) in naïve group 1 pulmonary hypertension.

DETAILED DESCRIPTION:
Introduction:

Pulmonary hypertension is pathophysiological condition defined as increases of mean pulmonary artery pressure above 20 mmHg as assessed by right heart catheterization (RHC) (1).

As pulmonary hypertension has a variety of causes with different clinical presentations and characteristics; it is classified into five clinical groups (2):

* Group 1 and also called pulmonary arterial hypertension group.
* Group 2 due to left sided heart diseases.
* Group 3 caused by chronic lung diseases and hypoxemia.
* Group 4 caused by chronic pulmonary artery occlusions.
* Group 5 that has unclear and multifactorial causes. Although group 1 less common; it is carrying significant clinical importance as early detection can improve the patient's outcome through providing them the available vasodilator medications.

To diagnose patient in group 1 PH, the patient should have RHC (3) to obtain the definite hemodynamic before starting treatment as advised by PH guidelines, however RHC is invasive and expensive procedure and carrying some bad drawback (4).

Transthoracic echocardiography is less expensive, non-invasive and nonhazardous procedure and commonly provide significant parameters before RHC (5).

several echocardiographic indices correlate significantly with RHC hemodynamic, as peak tricuspid regurgitation velocity , right ventricular outflow acceleration time, peak early pulmonary regurgitation velocity , peak late pulmonary regurgitation velocity, tricuspid regurgitation time velocity integral ,and tricuspid annulus tissue Doppler image velocities. Most of these parameters used individually to echocardiographic diagnose PH, however little data available to integrate them together to echocardiographic diagnose PH in group1; integrations of theses parameters might improve PH diagnosis As pulmonary arterial hypertension is Patho biological disease, and affecting small pulmonary arteries and arterioles, the pathologic pattern of vascular lesions is characterized by intimal hyperplasia, medial thickness, plexiform lesions, and thrombosis in situ, and is caused by increased migration and proliferation of smooth muscle cells (SMCs) and adventitial fibroblasts, abnormal endothelial cell proliferation, and impaired apoptosis (6).

several biomarkers play significant role in pathogenesis and prognosis of the diseases, serum uric acid (7,8) and serum troponin (9) may increase in PH and may affecting the clinical severity however further studies needed to confirm this .

Also micro RNA new marker of assessing cardiovascular diseases , may have role in assessing group 1 pulmonary hypertension(10).

ELIGIBILITY:
Inclusion Criteria:

1. Age>18 years old
2. Patient diagnosed as group 1 PH.

Exclusion Criteria:

1. Age under 18 years.
2. Unwilling or unable to sign the informed consent form.
3. Hemodynamically unstable condition requiring inotropic or vasoactive drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of echocardiographic indices in Group 1 pulmonary hypertension | baseline
  All trans thoracic echocardiographic indices will be measured:
  peak tricuspid regurgitation velocity (m/s). right ventricular outflow acceleration time (msec). peak early pulmonary regurgitation velocity (m/s). peak late pulmonary regurgitation velocity (m/s) . tricuspid regurgitation time velocity integral (m/s). tricuspid annulus tissue Doppler image . right ventricle morphology and functions. left ventricle morphology and functions.
Evaluation of serum troponin level in Group 1 pulmonary hypertension | baseline
  Blood samples from pulmonary circulation will be obtained for troponin level
Evaluation of serum uric acid in Group 1 pulmonary hypertension | baseline
  Blood samples from pulmonary circulation will be obtained for serum uric acid.

SECONDARY OUTCOMES:
Evaluation of mRNA level in Group 1 pulmonary hypertension | baseline
  Blood samples from pulmonary circulation will be obtained for mRNA level

REFERENCES:
- [Background] Simonneau G, Montani D, Celermajer DS, Denton CP, Gatzoulis MA, Krowka M, Williams PG, Souza R. Haemodynamic definitions and updated clinical classification of pulmonary hypertension. Eur Respir J. 2019 Jan 24;53(1):1801913. doi: 10.1183/13993003.01913-2018. Print 2019 Jan. PMID 30545968
- [Background] Simonneau G, Galie N, Rubin LJ, Langleben D, Seeger W, Domenighetti G, Gibbs S, Lebrec D, Speich R, Beghetti M, Rich S, Fishman A. Clinical classification of pulmonary hypertension. J Am Coll Cardiol. 2004 Jun 16;43(12 Suppl S):5S-12S. doi: 10.1016/j.jacc.2004.02.037. PMID 15194173
- [Background] Voelkel NF, Gomez-Arroyo J, Abbate A, Bogaard HJ. Mechanisms of right heart failure-A work in progress and a plea for failure prevention. Pulm Circ. 2013 Jan;3(1):137-43. doi: 10.4103/2045-8932.109957. No abstract available. PMID 23662190
- [Background] Voelkel NF, Tuder RM. Cellular and molecular biology of vascular smooth muscle cells in pulmonary hypertension. Pulm Pharmacol Ther. 1997 Oct-Dec;10(5-6):231-41. doi: 10.1006/pupt.1998.0100. No abstract available. PMID 9778486
- [Background] Bendayan D, Shitrit D, Ygla M, Huerta M, Fink G, Kramer MR. Hyperuricemia as a prognostic factor in pulmonary arterial hypertension. Respir Med. 2003 Feb;97(2):130-3. doi: 10.1053/rmed.2003.1440. PMID 12587962
- [Background] Filusch A, Giannitsis E, Katus HA, Meyer FJ. High-sensitive troponin T: a novel biomarker for prognosis and disease severity in patients with pulmonary arterial hypertension. Clin Sci (Lond). 2010 Jun 2;119(5):207-13. doi: 10.1042/CS20100014. PMID 20412051
- [Background] Crosswhite P, Sun Z. Nitric oxide, oxidative stress and inflammation in pulmonary arterial hypertension. J Hypertens. 2010 Feb;28(2):201-12. doi: 10.1097/HJH.0b013e328332bcdb. PMID 20051913